CLINICAL TRIAL: NCT02474225
Title: Intraocular Pressure Change Following Intravitreal Injection of Anti-vascular Endothelial Growth Factor Agent
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Weerawat Kiddee, Asst. Prof., Prince of Songkla University
Other Study IDs: EC-56-168-02-4-2
Record Dates: First submitted 2015-06-11; First posted 2015-06-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Intraocular Pressure
Keywords: intraocular pressure; intravitreal
MeSH Terms: interventions — Intravitreal Injections; Bevacizumab; Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Intravitreal injection (bevacizumab or ranibizumab) — The intravitreal anti-vascular endothelial growth factor agent of 0.1 ml of bevacizumab (2.5 mg/0.1 ml) or ranibizumab (1 mg/0.1 ml)
  Other Names: anti-vascular endothelial growth factor agent

SUMMARY:
The introduction of additional fluid into the vitreous cavity by intravitreal therapy would be expected to cause an immediate rise in the intraocular pressure. This transient, short-term intraocular pressure elevation (lasting up to 30 minutes) after intravitreal anti-vascular endothelial growth factor therapy has been well describe. The investigators aim to study the prevalence of the sustained intraocular pressure elevation associated with intravitreal injection of anti-vascular endothelial growth factor agents.

DETAILED DESCRIPTION:
Intravitreal injections of anti-vascular endothelial growth factor agents are commonly used to treat a variety of retinal and choroidal neovascular diseases. The introduction of additional fluid into the vitreous cavity by intravitreal therapy would be expected to cause an immediate rise in the intraocular pressure.

Although there is one study showed no significant changes in the intraocular pressure many retrospective studies showed the impacts on the intraocular pressure elevation. The investigators aim to prospective evaluate the intraocular pressure change in non-glaucomatous patients receiving an intravitreal anti-vascular endothelial growth factor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to receive intravitreal injection of anti-vascular endothelial growth factor agent (either bevacizumab or ranibizumab), and
* Age of 18-85 year-old, and
* Initial intraocular pressure < 21 mmHg

Exclusion Criteria:

* Diagnosis of open angle, or
* Diagnosis of angle-closure glaucoma, or
* Diagnosis of glaucoma suspect (intraocular pressure > 21 mmHg on 2-consecutive visit and/or cup to disc ratio > 0.5) , or
* Currently receive systemic beta-blocker
* Previously received intravitreal injection of anti-vascular endothelial growth factor agent
* Previously received intravitreal injection of steroid or gancyclovir
* Current use of steroid eye drop
* Any ocular surface disease preclude a reliable intraocular pressure measurement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients scheduled to receive intravitreal injection of anti-vascular endothelial growth factor agent (either bevacizumab or ranibizumab) and were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in intraocular pressure | 6-month after injection
  intraocular pressure change at 6-month after injection

SECONDARY OUTCOMES:
Number of anti-glaucoma used | 6-month
  Start anti-glaucoma If there is an increase in intraocular pressure over the target IOP

CONTACTS AND LOCATIONS:
Overall Officials: Asst.Prof.Weerawat Kiddee, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Weerawat Kiddee, Hat Yai, Changwat Songkhla, Thailand